CLINICAL TRIAL: NCT04558164
Title: Network-targeted Theta-burst Stimulation for Episodic Memory Improvement in Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nanthia Suthana, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-001417; R01AG068317 (NIH)
Record Dates: First submitted 2020-09-04; First posted 2020-09-22 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Dysfunction; Memory Disorders in Old Age
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TBS (Experimental): Theta burst stimulation (TBS) will be delivered at 100% of motor threshold (MT).
  Interventions: Device: Active Theta Burst Stimulation
- Sham TBS (Sham Comparator): Sham stimulation will be delivered at 0% of motor threshold (MT), with all other parameters matching the active TBS condition.
  Interventions: Device: Sham Theta Burst Stimulation

INTERVENTIONS:
Device: Active Theta Burst Stimulation — Theta burst transcranial magnetic stimulation (TBS) will be delivered at 80-100% of motor threshold (MT).
  Arms: Active TBS
Device: Sham Theta Burst Stimulation — Sham stimulation will be delivered at 0-10% of motor threshold (MT), with all other parameters matching the active TBS condition.
  Arms: Sham TBS

SUMMARY:
The purpose of this study is to see if stimulation of the brain can improve memory. The investigators will use a device called transcranial magnetic stimulation that can stimulate and activate a specific part of the brain that is important for memory. The study will enroll MCI subjects and subjects with subjective memory complaints who will be randomly assigned to receive active or sham brain stimulation. 'Blinded' or 'sham-controlled' means that the subject will not know whether the treatment they receive is the active treatment or the non-active stimulation. In the 'sham' condition, the stimulator will turn on but will not actually be stimulating the target brain region.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate in the study
* 55-100 years of age
* Right-handedness
* In good general health
* Living independently
* Subjective memory complaints (self-report and positive score on MFQ)
* Katz ADL scale and Lawton iADL scale: We will review scores on a case-by-case basis if they did not score 100%. We will exclude if the scores show impairment in ADLs that suggests problems with independent functioning due to cognitive impairment.
* MMSE score > 24
* PHQ Depression score =< 7
* Ability to read, write, and speak English fluently
* Diagnosis of mild neurocognitive disorder according to DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) criteria. Participants with subjective memory complaints without an aMCI diagnosis will be reviewed on a case-by-case basis based on neuropsychological scores. Participants scoring a raw score of 0 or 3 standard deviations below normative expectations on the long delay recall in two or more of the three tasks (BVMT-R, RCFT, and CVLT-III) will be excluded.
* No change in use of psychotropic medication for treatment of depression, anxiety, ADHS or psychosis 1 month prior and during the study.

Screening diagnostic criteria for aMCI will be subjective memory complaints, intact instrumental and basic activities of daily living (Smith et al., 1996), PHQ, MMSE, BVMT-R (25-minute delay), CVLT-II (20-minute delay), Rey-Osterrieth Complex Figure Task (30-minute delay). Baseline assessments will include neuropsychological testing of all study subjects.

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Diagnosis of dementia
* Active major medical, psychiatric, or neurologic disorder associated with neurocognitive impairment
* History of alcohol or substance abuse
* Recent (< 6 months) alcohol or substance abuse (excluding nicotine or caffeine)
* History of stroke (if the stroke in our judgment is related to the memory problem), traumatic brain injury with loss of consciousness, or other neurologic disorder (e.g., epilepsy, Huntington's disease, Parkinson's disease)
* Non-English speaking participants
* Not right handed based on self-report or evaluation based on a standard report
* Has received TMS before (not TMS naïve)
* Poorly controlled hypertension or cardiovascular disease
* Current enrollment in a memory-enhancement study or course
* Contraindication to TMS or MRI including claustrophobia, metal in body, surgery within 60 days, certain implants, or previous abnormal MRI results.
* scanning facial tattoos is okay if safe with MRI
* is taking:

  * anticholinergic medication (e.g., Detrol, Cogentin);
  * sedating antihistamine (e.g., Benadryl);
  * any drug that has significant anticholinergic or antihistaminic side effects (e.g., tricyclic antidepressant medications, Remeron).
  * benzodiazepines. While not a strict rule out, this will be decided on a case-by-case basis depending on the dose.

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Verbal recall performance change | Baseline: Day 2; During stimulation: Day 3, Day 7, Day 12, Day 17; Follow-up appointments: Day 18, Day 19, Day 20.
  Verbal memory will be measured using a free recall task where participants learn a list of everyday words and are asked to recall as many words as they can remember after a period of distraction. Proportion of recollected words will be used to quantify memory performance changes.
Object recognition memory performance change | Baseline: Day 2; During stimulation: Day 3, Day 7, Day 12, Day 17; Follow-up appointments: Day 18, Day 19, Day 20.
  Object memory will be measured using an recognition task where participants view photos of everyday objects and are asked to identify them as OLD or NEW during a memory test wherein unseen novel objects and very similar but new photos of identical objects are shown. Recollection and discrimination index will be used to quantify memory performance changes.
Associative memory performance change | Baseline: Day 2; During stimulation: Day 3, Day 7, Day 12, Day 17; Follow-up appointments: Day 18, Day 19, Day 20.
  Associative memory will be tested using the Face Name Memory Test wherein participants are shown faces and associated names. Participants are then shown faces only and asked to recall the associated name.

SECONDARY OUTCOMES:
Resting state fMRI functional connectivity | Baseline (Day 2) before the first treatment and after the last treatment (Day 17)
  Resting state fMRI activity will be measured before the first and after the last TBS treatment
EEG activity | During treatment (Days 3, 7 and 12), after the last treatment (Day 17), and 2 month follow-up session (Day 20)
  EEG functional connectivity with stimulated region and medial temporal source localized power in the theta band will be recorded during a resting period as well as during the treatment itself both before and after treatments

CONTACTS AND LOCATIONS:
Overall Officials: Nanthia Suthana, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The data collected for this research represent a valuable resource to the scientific community, and the PIs will make them accessible to others, while respecting the special needs for confidentiality. All data will be anonymized before being provided to the scientific community. Researchers can also request access to the data under collaborative and co-authorship agreements prior to the end of the funding period or before publication. The results from the proposed project will also be shared at scientific meetings (local, national and international) as well via published manuscripts.
Time Frame: All data will be provided by the time publication occurs or when the proposed funding period has ended.
Access Criteria: Researchers can request access to the data under collaborative and co-authorship agreements prior to the end of the funding period or before publication.